CLINICAL TRIAL: NCT03825523
Title: Impact of the Timing of Antiretroviral Therapy Initiation (Immediate Versus Early) on the Mortality Rate of HIV/AIDS Patients Hospitalized With an Opportunistic Disease
Brief Title: Immediate ART in Subjects With Opportunistic Diseases
Acronym: TARi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustavo Reyes-Teran (Other Government)
Responsible Party: Sponsor-Investigator, Gustavo Reyes-Teran, Principal Investigator, Centro de Investigación en. Enfermedades Infecciosas, Mexico
Organization: Centro de Investigación en. Enfermedades Infecciosas, Mexico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C09-18
Record Dates: First submitted 2019-01-18; First posted 2019-01-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HIV/AIDS; ANTIRETROVIRAL TREATMENT
Keywords: HIV/AIDS; ART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Stratified randomization will be generated by an electronic system, in blocks of 6 and 8, and a 1:1 ratio, according to the CD4+ T cell count.
  Group A: Immediate treatment (iART). Start ART within 48 hours of admission and hospitalization; Group B: Conventional treatment (cART). Start the ART once the opportunistic infection is under control at the discretion of infectious disease specialist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Immediate treatment (iART) (Experimental): Other: time to start the ART within 48 hours of admission to hospitalization
  Interventions: Other: iART
- Group B Conventional treatment (cART) (Active Comparator): Other: time to start the ART, after the opportunistic disease has been controlled, at the discretion of infectious disease specialist.
  Interventions: Other: cART

INTERVENTIONS:
Other: iART — After group assignment, ART will be started within the first 48 hours after admission to the hospital. ART regimen will be decided according to each subject´s the clinical characteristics
  Arms: Group A Immediate treatment (iART)
Other: cART — After group assignment, ART is started at the discretion of the attending physician. ART regimen will be decided according to each subject´s the clinical characteristics
  Arms: Group B Conventional treatment (cART)

SUMMARY:
The aim of this study is to compare the clinical response and mortality rate by an opportunistic disease in HIV-infected individuals who start immediate versus conventional antiretroviral therapy.

Immediate ART (iART) is defined as starting antiretroviral therapy in the first 48 hours after the hospitalization.

Conventional ART (cART) is defined as starting antiretroviral therapy once the opportunistic infection is under control at the discretion of infectious disease specialist.

DETAILED DESCRIPTION:
Sample size was calculated using formula, of difference in proportions formula using a beta of 0.1, alpha of 0.05 and an expected difference in mortality of 20%, The sample size is 225 subjects in each group. Informed consent will be obtained. Patients will be allocated to each group (iART or cART) after randomization stratified by the CD4+ T cell count (less or more than 50 cells/mm3).

Plasma viral load and CD4+ T cell count will be measured at study entry and at weeks 2, 4, 12, 24 and 48 after ART initiation. Clinical outcomes will be: mortality at 4, 12, 24, and 48 weeks, length of hospitalization (measured in days), clinical and microbiological cure of the opportunistic disease, incidence and severity of immune reconstitution of inflammatory syndrome (IRIS), and adverse drug reactions and interactions.

Once 50% of the sample size has completed 30 days of follow-up, a preliminary analysis will be conducted to assess safety and efficacy of iART; if differences in the mortality are observed, the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Time from admission to study entry: less than 48 hours
* Confirmed HIV diagnosis or high probability of HIV infection based on a positive HIV rapid test
* Having an opportunistic disease
* Subjects must be naïve to ART or have failed their first or second ART regimen or must have abandoned ART for more than 3 months

Exclusion Criteria:

* Meningitis due to Cryptococcus spp. or for M. tuberculosis
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Compare mortality rates betweeno two groups according to the timing of ART initiation: immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART)

SECONDARY OUTCOMES:
Assess survival rates | 90 days since starting antiretroviral therapy (ART)
  Compare the survival rate of HIV-infected patients on immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART)
Assess survival rates | 180 days since starting antiretroviral therapy (ART)
  Compare the survival rate of HIV-infected patients on immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART)
Assess survival rates | 360 days since starting antiretroviral therapy (ART)
  Compare the survival rate of HIV-infected patients on immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART)
Length of stay | 1 year
  Compare length of hospitalization between both groups
Asses survival rates by the CD4 count | 90 days
  Compare the survival rate of HIV-infected patients on immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART) stratified by CD4+ T cell count at study entry
Asses survival rates by the CD4 count | 180 days
  Compare the survival rate of HIV-infected patients on immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART) stratified by CD4+ T cell count at study entry
Asses survival rates by the CD4 count | 360 days
  Compare the survival rate of HIV-infected patients on immediate antiretroviral therapy (iART) versus conventional antiretroviral therapy (cART) stratified by CD4+ T cell count at study entry
Viral load | 90 days
  Measure the baseline plasma viral load and evaluate its dynamics after ART initiation in both groups
Viral load | 180 days
  Measure the baseline plasma viral load and evaluate its dynamics after ART initiation in both groups
Viral load | 360 days
  Measure the baseline plasma viral load and evaluate its dynamics after ART initiation in both groups
CD4 T cell counts | 90 days
  Measure CD4+ T cell counts, and evaluate its dynamics after ART initiation in both groups
CD4 T cell counts | 180 days
  Measure CD4+ T cell counts, and evaluate its dynamics after ART initiation in both groups
CD4 T cell counts | 360 days
  Measure CD4+ T cell counts, and evaluate its dynamics after ART initiation in both groups
IRIS | 48 weeks
  Determine the incidence and severity of IRIS. Severity will be classified as mild or life threatening
Adverse reactions | 48 weeks
  Describe ART-related adverse events, and drug interactions

CONTACTS AND LOCATIONS:
Overall Officials: GUSTAVO MD REYES-TERÁN, M.D., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Centro de Investigacion en Enfermedades Infecciosas, México, State of Mexico, Mexico